CLINICAL TRIAL: NCT07336095
Title: Effect of Oral Melatonin Versus Oral Midazolam as a Premedication in Children Undergoing Tonsillectomy
Brief Title: Melatonin vs Midazolam in Children Undergoing Tonsillectomy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Wael Sayed El Gharabawy, assisstant professor of anesthesia, intensive care, and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MS 206/2025
Record Dates: First submitted 2025-11-24; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Emergence Delirium, Anesthesia; Child; Anxiety; Midazolam Premedication; Melatonin Bioavailability; Tonsillectomy
Keywords: melatonin, midazolam, anxiety, children, tonsillectomy
MeSH Terms: conditions — Emergence Delirium; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Melatonin group (Group M) (Active Comparator): All patients will be subjected to a thorough medical history, physical examination, routine preoperative investigations will be done to all children including laboratory investigations as (complete blood picture, bleeding time, prothrombin time and partial thromboplastin time). Age, weight, and sex will be recorded.
  One hour before sedation, children will be transported to an isolated recovery room near the operation room. Parental presence will be allowed throughout sedation and post sedation period. Patients will be randomly assigned to three groups first group(M group) will receive 0.3 mg per kg oral melatonin in 10 ml Dextrose 10% 45 min before surgery )Maximum dose 10mg). Assessment of sedation and anxiolysis 30 min after the drug administration using Ramsay sedation scale.
  Interventions: Drug: Melatonin group
- Midazolam group (Group D) (Sham Comparator): All patients will be subjected to a thorough medical history, physical examination, routine preoperative investigations will be done to all children including laboratory investigations as (complete blood picture, bleeding time, prothrombin time and partial thromboplastin time). Age, weight, and sex will be recorded. One hour before sedation, children will be transported to an isolated recovery room near the operation room. Parental presence will be allowed throughout sedation and post sedation period. Patients will be randomly assigned to three groups first group(M group) will receive 0.3 mg per kg oral midazolam in 10 ml Dextrose 10% 45 min before surgery )Maximum dose 10mg). Assessment of sedation and anxiolysis 30 min after the drug administration using Ramsay sedation scale.
  Interventions: Drug: Midazolam group
- placebo group (Group C) (Placebo Comparator): All patients will be subjected to a thorough medical history, physical examination, routine preoperative investigations will be done to all children including laboratory investigations as (complete blood picture, bleeding time, prothrombin time and partial thromboplastin time). Age, weight, and sex will be recorded. One hour before sedation, children will be transported to an isolated recovery room near the operation room. Parental presence will be allowed throughout sedation and post sedation period. Patients will will receive 10 ml pure oral Dextrose 10% 45 min before surgery. Assessment of sedation and anxiolysis 30 min after the drug administration using Ramsay sedation scale.
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Melatonin group — All patients will be subjected to a thorough medical history, physical examination, and routine preoperative investigations will be done to all children, including laboratory investigations (complete blood picture, bleeding time, prothrombin time, and partial thromboplastin time). Age, weight, and sex will be recorded.
  One hour before sedation, children will be transported to an isolated recovery room near the operating room. Parental presence will be allowed throughout the sedation and post-sedation period.
  Patients will receive 0.3 mg per kg oral melatonin in 10 ml Dextrose 10% 45 min before surgery (Maximum dose 10mg). Assessment of sedation and anxiolysis 30 min after the drug administration using Ramsay sedation scale.
  Arms: Melatonin group (Group M)
Drug: Midazolam group — All patients will be subjected to a thorough medical history, physical examination, and routine preoperative investigations will be done to all children, including laboratory investigations (complete blood picture, bleeding time, prothrombin time, and partial thromboplastin time). Age, weight, and sex will be recorded.
  One hour before sedation, children will be transported to an isolated recovery room near the operating room. Parental presence will be allowed throughout the sedation and post-sedation period.
  Patients will receive 0.3 mg per kg oral midazolam in 10 ml Dextrose 10% 45 min before surgery (Maximum dose 10mg). Assessment of sedation and anxiolysis 30 min after the drug administration using Ramsay sedation scale.
  Arms: Midazolam group (Group D)
Drug: Control group — All patients will be subjected to a thorough medical history, physical examination, and routine preoperative investigations will be done to all children, including laboratory investigations (complete blood picture, bleeding time, prothrombin time, and partial thromboplastin time). Age, weight, and sex will be recorded.
  One hour before sedation, children will be transported to an isolated recovery room near the operating room. Parental presence will be allowed throughout the sedation and post-sedation period.
  Patients will receive 10 ml pure oral Dextrose 10% 45 min before surgery. Assessment of sedation and anxiolysis 30 min after the drug administration using Ramsay sedation scale.
  Arms: placebo group (Group C)

SUMMARY:
Used as a premedication to decrease anxiety (Caumo et al., 2007). Midazolam, though has several drawbacks (McCann and Kain, 2001). Hence, an alternative premedication to midazolam will definitely have a widespread appeal.

Melatonin is a hormone secreted by the pineal gland. Melatonin is different from benzodiazepines and their derivatives in that it exerts a promoting effect on sleep by amplifying day/night differences in alertness and sleep quality and displaying a modest sleep-inducing effect, quite mild as compared to that seen with benzodiazepines (Ahmad et al., 2007). Melatonin has also been reported to cause preoperative anxiolysis and an increase in levels of sedation without impairing orientation (Naguib and Samarkandi, 2000). Hence, the aim of this study is to compare the effect of oral melatonin and oral midazolam on preoperative anxiety.

Emergence delirium (ED) was first described in the literature in the early 1960s. Although often used interchangeably with emergence agitation, it is defined as a temporary dissociated state of consciousness after discontinuation of anesthesia. The characteristics that make up ED include irritability, inconsolable crying, distress and inability to cooperate (Reduque and Verghese, 2013).

Midazolam is the most prescribed oral premedication in the preoperative setting. Its benefits include preoperative anxiolysis, amnesia, relatively rapid onset and short duration of action. Although most children have anxiolysis with midazolam, up to 29% may display a paradoxical agitation response (Shin et al., 2013).

Oral melatonin doses up to 0.4 mg/kg (maximum 20 mg) are effective in reducing ED in children (age 3-7 years) (Kain et al., 2009).

AIM OF THE WORK The study aims to compare the effects of oral melatonin and oral midazolam on preoperative anxiety as a premedication in children undergoing tonsillectomy.

DETAILED DESCRIPTION:
Preoperative anxiety is a common and significant concern in pediatric patients undergoing surgery. Anxiety is defined as a feeling of apprehension, fear, or uneasiness about an anticipated event, and in the surgical setting, it arises primarily from the fear of separation from parents, unfamiliar environments, painful stimuli, and the unknown nature of the procedure itself (Kain et al., 2006). Studies estimate that up to 60-70% of children experience substantial preoperative anxiety, with younger children, those with shy temperaments, and those undergoing repeated surgeries being at higher risk (Chow et al., 2016).

Causes and Contributing Factors Several factors contribute to heightened anxiety in children before surgery. These include developmental stage, previous hospitalizations, parental anxiety levels, lack of adequate preparation or information, and the presence of unfamiliar medical personnel (Fortier et al., 2010). Children aged between 1 and 5 years are especially vulnerable due to their limited coping mechanisms and fear of separation. A child's temperament, such as shyness or behavioral inhibition, also influences anxiety levels (Davidson et al., 2006).

Clinical Implications of Preoperative Anxiety Unmanaged preoperative anxiety has both immediate and long-term consequences. It can lead to increased distress during induction of anesthesia, higher requirements for anesthetic agents, postoperative pain, emergence delirium, and delayed recovery (Kain et al., 2004). Moreover, there is a correlation between preoperative anxiety and the development of postoperative maladaptive behaviors such as nightmares, bedwetting, aggression, and eating disturbances (Yuki and Daaboul, 2011) Assessment of Preoperative Anxiety Quantifying anxiety in children is essential for guiding intervention. Several validated tools are available, including the Modified Yale Preoperative Anxiety Scale (m-YPAS), which evaluates behaviors like activity level, vocalization, emotional expressivity, and use of parents. This scale is reliable in assessing anxiety levels during the preoperative period (Ramkisson, 2019).

Management Strategies Preoperative anxiety in children is a multifaceted problem that significantly affects surgical outcomes. Early identification and appropriate interventions, both behavioral and pharmacological, can reduce anxiety levels, improve compliance, and contribute to better perioperative experiences (Matthias and Samarasekera, 2012).

Management of preoperative anxiety in children includes both pharmacological and non-pharmacological methods. Non-drug approaches include parental presence during induction, behavioral interventions (e.g., distraction, play therapy, video games), and preoperative education. Pharmacological agents such as midazolam and melatonin are also widely used for anxiolysis. A multimodal approach is often the most effective (Agbayani et al., 2020).

PREOPERATIVE SEDATION AND PREMEDICATION IN PEDIATRICS T The goal of preoperative sedation and premedication is to reduce anxiety, facilitate smooth induction of anesthesia, decrease psychological trauma, and improve the overall perioperative experience. Children are particularly vulnerable to preoperative stress, making the selection of safe and effective premedication essential (Dave, 2019).

Premedication in children has evolved significantly over the past decades. Initially, sedatives such as chloral hydrate and opioids were used, but concerns regarding safety and postoperative respiratory depression shifted focus toward benzodiazepines and other safer agents. In recent years, natural compounds like melatonin have emerged as alternatives to synthetic sedatives (Beckman et al., 2017).

Classification of Sedation Techniques

Sedation techniques can be classified as:

Pharmacological Includes benzodiazepines (e.g., midazolam), alpha-2 agonists (e.g., clonidine, dexmedetomidine), antihistamines, and melatonin (Taghizadeh et al., 2015).

Non-pharmacological Includes parental presence, audiovisual distraction (e.g., cartoons), hypnosis, cognitive behavioral therapy, and music therapy (Kulakaç and Ustuner Top, 2025).

Routes of Administration

Premedication can be administered via various routes depending on the agent and patient preference:

* Oral: Most commonly used; easy to administer and well accepted.
* Intranasal: Provides rapid onset; used for drugs like midazolam and dexmedetomidine (Yuen et al., 2008, Sheta et al., 2014).
* Intramuscular: Less favored due to pain and fear.
* Rectal: Occasionally used, especially in uncooperative children.
* Sublingual and Buccal: Emerging routes for faster absorption without invasive administration (Szczeklik and Fronczek, 2021).

Criteria for Ideal Premedication

An ideal premedication agent in pediatrics should:

* Be effective in reducing anxiety and facilitating separation
* Have a rapid onset and short duration
* Be easy to administer and acceptable by the child
* Have minimal side effects
* Not delay recovery or discharge
* Commonly Used Agents (Dave, 2019) Table 1: Ideal Premedication Criteria and Commonly Used Agents in Pediatrics (Dave, 2019).

Premedication reduces anxiety, minimizes crying during separation and induction, and can improve compliance. The choice of agent depends on child characteristics, surgery type, and institutional protocols. Oral midazolam remains the gold standard, but melatonin is increasingly favored for its natural origin and fewer adverse effects (Isik et al., 2008).

Preoperative sedation and premedication are crucial in pediatric anesthesia. A tailored approach using both pharmacologic and behavioral strategies ensures optimal outcomes. The emergence of agents like melatonin is promising, particularly in cases where minimizing side effects is a priority (Rana et al., 2024).

General Contraindications to Preoperative Sedation in Pediatrics While preoperative sedation is beneficial in reducing anxiety and facilitating smooth induction, it is not universally safe for all pediatric patients. Several clinical scenarios warrant caution or complete avoidance of sedative premedication due to the risk of adverse effects or worsening of the underlying condition (Yang et al., 2022).

1. Absolute Contraindications

   These are conditions where sedation is clearly contraindicated:
   * Severe airway obstruction (e.g., large tonsils with obstructive sleep apnea): Sedation may worsen airway collapse (Malviya et al., 2004).
   * Unstable cardiopulmonary status: Sedatives can depress respiratory or cardiac function (Jang and Kim, 2024)
   * Raised intracranial pressure: Certain sedatives (e.g., ketamine) may increase cerebral blood flow and pressure (Jang and Kim, 2024)
   * Known hypersensitivity or allergy to the sedative agent (Hertzog et al., 2019).
   * Lack of appropriate monitoring equipment or trained personnel for managing airway and emergencies (Pediatrics et al., 2006).
2. Relative Contraindications

   These require careful assessment and individualized risk-benefit analysis:
   * Severe hepatic or renal impairment: Affects metabolism and clearance of most sedatives.
   * Neurologic disorders (e.g., epilepsy): Some sedatives may lower seizure threshold.
   * Previous adverse reaction to sedation or paradoxical agitation.
   * Delayed gastric emptying or full stomach: Increases aspiration risk during deep sedation.
   * Parental refusal or lack of consent: Ethical and legal contraindication (Friedman, 2011) (Battaglini and De Rosa, 2024).
3. Caution in Certain Populations

   * Infants under 6 months: Immature organ systems may increase risk of apnea and bradycardia.
   * Children with developmental delay or autism: May have atypical responses or require adjusted dosing.
   * Severe malnutrition or dehydration: Alters drug distribution and clearance (Horeczko and Mahmoud, 2021).

MIDAZOLAM M idazolam is a water-soluble benzodiazepine derivative used widely in pediatric anesthesia for preoperative anxiolysis, sedation, and as an induction adjunct. It was first synthesized in 1976 and introduced clinically due to its rapid onset, short duration, and relative safety compared to diazepam. It functions primarily as a positive allosteric modulator at GABA-A receptors, enhancing the effect of endogenous GABA by increasing the frequency of chloride channel opening, resulting in hyperpolarization and decreased neuronal excitability (Khurmi et al., 2017).

Pharmacodynamics and Pharmacokinetics Midazolam exhibits dose-dependent effects, ranging from anxiolysis at low doses to hypnosis and amnesia at higher doses (Hong, 2022). It is unique among benzodiazepines for its pH-dependent ring structure: in acidic solutions, it is water-soluble, but at physiological pH, it becomes lipophilic, facilitating rapid brain uptake. Its volume of distribution in children is larger than in adults, and its half-life ranges from 1.5 to 3 hours in healthy pediatric patients. In neonates and infants, the half-life may be prolonged due to immature liver enzyme systems (Coté and Wilson, 2008).

Midazolam undergoes hepatic metabolism via the CYP3A4 enzyme, producing an active metabolite, 1-hydroxymidazolam, which contributes to its sedative effects but is less potent. Renal excretion eliminates both the parent drug and its metabolites. Thus, caution is required in patients with hepatic or renal dysfunction (Flores-Pérez et al., 2023).

Figure 1: Midazolam Metabolism and Mechanism of Action (Smith et al., 1981, Reves et al., 1985) Routes of Administration

* Oral (0.5 mg/kg): Most commonly used for pediatric premedication. It has a relatively rapid onset (15-30 minutes) and acceptable taste when mixed with juice (Dowdy et al., 2023).
* Intranasal (0.2 mg/kg): Offers rapid absorption through the nasal mucosa, particularly useful in uncooperative children, with onset in 5-10 minutes (Shah et al., 2024).
* Intravenous (0.05-0.1 mg/kg): Preferred for titratable and immediate sedation in procedural or intraoperative use (Necula et al., 2025).
* Intramuscular (0.1-0.15 mg/kg): Less favored due to pain on injection and variable absorption, but still used when IV access is unavailable (Coté and Wilson, 2008).
* Rectal or Buccal: Employed particularly in seizure emergencies or in children where IV access is not feasible (Coté and Wilson, 2008).

Clinical Applications

Midazolam is used extensively in pediatric anesthesia:

* Premedication before induction.
* Procedural sedation for imaging, endoscopy, or minor surgeries.
* Seizure control in acute settings (especially intranasal or buccal).
* Induction adjunct for children undergoing balanced anesthesia (Lethin et al., 2023) (Jacqz-Aigrain and Choonara, 2021).

It reduces separation anxiety during parental handover, improves mask acceptance, and provides anterograde amnesia, thus minimizing traumatic memory formation. It is often combined with ketamine or opioids to enhance sedation and analgesia (Coté and Wilson, 2008).

Safety and Side Effects

Though generally safe when used appropriately, midazolam is associated with several potential adverse effects:

* Respiratory depression, especially in high doses or when combined with opioids or other CNS depressants (Coté and Wilson, 2008).
* Paradoxical reactions such as agitation, disinhibition, or restlessness occur in 1-15% of children, and are more common with higher doses or rapid IV administration (Peter et al., 2024).
* Delayed recovery or a "hangover effect" may occur, especially in neonates or those with hepatic or renal dysfunction due to prolonged half-life (Karunarathna et al., 2025)
* Hypotension, although uncommon, can occur particularly when midazolam is used with other sedatives or in hemodynamically unstable patients (Cappellini et al., 2024).
* Therefore, continuous monitoring of oxygen saturation, respiratory rate, and sedation depth is essential in all children receiving midazolam (Coté and Wilson, 2008) (Peter et al., 2024).

Evidence-Based Effectiveness Studies have shown midazolam to be superior to placebo in reducing preoperative anxiety and improving induction quality. However, concerns about its cognitive effects, particularly amnesia and post-discharge behavior changes, have led researchers to explore alternative agents like melatonin (Samarkandi et al., 2005).

MELATONIN M elatonin is an indoleamine hormone synthesized from tryptophan in the pineal gland, especially in response to darkness. Beyond its role in regulating the circadian rhythm, melatonin has anxiolytic, hypnotic, analgesic, antioxidant, and anti-inflammatory effects that are increasingly utilized in pediatric anesthesia (Repova et al., 2022).

Pharmacology and Mechanism of Action Melatonin acts primarily on MT1 and MT2 G-protein coupled receptors, mainly located in the suprachiasmatic nucleus of the hypothalamus, hippocampus, and other CNS sites. MT1 promotes sleep induction, while MT2 regulates circadian phase shifts. Melatonin also modulates GABAergic, opioid, and nitric oxide pathways, explaining its multi-modal sedative and analgesic effects (Kurdi and Patel, 2013).

Figure 2: Pharmacology and Mechanism of Action (Sharma et al., 2015). Unlike benzodiazepines, melatonin does not cause respiratory depression, cognitive impairment, or addiction. Its elimination half-life is 30-60 minutes, but receptor interaction effects may last longer. It is metabolized in the liver by CYP1A2 and excreted as 6-sulfatoxymelatonin in urine (Beshir and Cook, 2021).

Pediatric Dosage and Administration

There is no universally agreed-upon pediatric dose, but commonly used regimens include:

* Oral: 0.2-0.5 mg/kg or fixed 3-6 mg, 30-60 minutes before anesthesia (Kurdi and Patel, 2013, Gitto et al., 2016).
* Sublingual: same dose, faster onset, ideal for children unable to swallow.
* Rectal or transdermal: explored in neonates or children with enteral access issues.

Melatonin is typically given 30-60 minutes before surgery, allowing sufficient time for peak serum levels (Naguib et al., 2007).

Clinical Applications in Pediatric Anesthesia

Melatonin provides effective premedication by:

* Reducing preoperative anxiety and stress-related cortisol levels
* Facilitating smoother parental separation
* Improving mask acceptance and IV cannula tolerance
* Reducing emergence delirium, particularly in preschoolers
* Supporting postoperative sleep and recovery quality (Chen et al., 2025). It has been studied as an alternative or adjunct to midazolam in various surgeries, including tonsillectomy, hernia repair, and dental procedures (Samarkandi et al., 2005).

Analgesic and Neuroprotective Effect Melatonin exerts antinociceptive effects by interacting with opioid receptors, calcium channels, and antioxidant pathways. It reduces the need for postoperative opioids and supports faster recovery. In neonates and preterm infants, melatonin shows neuroprotective potential in hypoxic-ischemic injury due to its antioxidant action (Gitto et al., 2016).

Safety Profile

Melatonin is remarkably well-tolerated:

* No respiratory or cardiovascular depression
* No memory impairment or behavioral dysregulation
* Low risk of hormonal interference with short-term use
* No dependency or withdrawal phenomena (Givler et al., 2023). Rare side effects include daytime drowsiness, headache, or mild mood changes, but these are infrequent at therapeutic doses (Coté and Wilson, 2008).

Table 2: Comparison between midazolam and melatonin (Peter et al., 2024) (Tordjman et al., 2017)

ELIGIBILITY:
Inclusion Criteria:

-ALL children with ASA class I and class II

Exclusion Criteria:

* chest infection
* Abnormal mental milestones.
* Children with any organ dysfunction.
* Allergies to any of the drugs used.
* Children with Obstructive sleep apnea.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of preoperative anxiety with oral melatonin vs oral midazolam as a premedication in Children Undergoing Tonsillectomy. | 30 minutes after giving the drug
  Assessment of sedation 30 min after the drug administration using Ramsay sedation scale.

SECONDARY OUTCOMES:
1. Effect of both drugs in reducing incidence of post operative emergence delerium | 24 hours afer the procedure
  Pediatric Anesthesia Emergence Delirium (PAED) Scale Score. The PAED scale consists of 5 criteria that are scored using a 5-point scale. The scores of each criterion are added to make a total score. The maximum achievable score is 20. A score of ≥10 has 64% sensitivity and 86% specificity for the diagnosis of ED. A score of >12 has 100% sensitivity and 94.5% specificity for the diagnosis of ED

IPD SHARING:
Plan to Share IPD: No